CLINICAL TRIAL: NCT03409835
Title: Effect of Ramosetron on Post-discharge Nausea and Vomiting in Patients Undergoing Gynecologic Surgery Through a Day-surgery Center
Brief Title: Effect of Ramosetron on Post-discharge Nausea and Vomiting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Hyo-Seok Na, Principle investigator, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PDNV
Record Dates: First submitted 2018-01-09; First posted 2018-01-24 (Actual); Last update posted 2018-04-20 (Actual); Status verified 2018-04

CONDITIONS: Hysteroscopy
MeSH Terms: interventions — ramosetron; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ramosetron (Experimental)
  Interventions: Drug: Ramosetron
- Control (Placebo Comparator)
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Ramosetron — Ramosetron 0.3 mg is administered after induction of general anesthesia.
  Arms: Ramosetron
Drug: Normal saline — Normal saline 2 ml is administered after induction of general anesthesia.
  Arms: Control

SUMMARY:
Nausea and vomiting after general anesthesia is one of the common anesthetic complications. If the patient is discharged from the hospital after surgery, proper treatment may be delayed or impossible if nausea or vomiting occurs. Thus, It is necessary to prevent these symptoms beforehand. Patients who underwent gynecologic surgery will be treated with prophylactic ramosetron to determine whether the frequency of nausea and vomiting is decreased when the patient returned home after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergo hysteroscopic surgery and are discharged on the day of surgery.

Exclusion Criteria:

* American Society of Anesthesiologists physical statue 3 or more
* Planned admission after surgery
* Intravenous anesthesia
* During chemotherapy
* Pregnancy or breastfeeding
* Abnormal liver or kidney function

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-02 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
The change in the occurrence of postoperative nausea | Postoperative 30 minute, 3 hour, 24 hour, and 48 hour
The change in the occurrence of postoperative vomiting | Postoperative 30 minute, 3 hour, 24 hour, and 48 hour

SECONDARY OUTCOMES:
The change of postoperative pain score | Postoperative 30 minute, 3 hour, 24 hour, and 48 hour
  Score range is from 0 to 10.
The change in the number of postoperative administration of rescue analgesic drug | Postoperative 30 minute and 3 hour
The change in the number of postoperative administration of rescue antiemetic drug | Postoperative 30 minute and 3 hour
The change of patient's satisfaction score | Postoperative 30 minute, 3 hour, 24 hour, and 48 hour
  Score range is from 0 to 10.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National Univ. Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea